CLINICAL TRIAL: NCT04947826
Title: A Randomized, Double-blinded, Controlled Phase II Study of Combination Therapy of HAIC (Hepatic Arterial Infusion Chemotherapy), HLX10 (PD-1 Antibody) and HLX04 (VEGF Antibody) Compared With HAIC and Placebo in Hepatocellular Carcinoma With Major Portal Vein Tumor Thrombosis
Brief Title: Combination Therapy of HAIC and HLX10 and HLX04 in HCC With Major Portal Vein Tumor Thrombosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HHH
Record Dates: First submitted 2021-06-18; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Hepatocellular Carcinoma With Major Portal Vein Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC + HLX10 + HLX04 (Experimental): HAIC: FOLFOX, q3w, up to 8 times; HLX10: 4.5mg/kg, iv, q3w, up to 2 years; HLX04: 15.0mg/kg, iv, q3w, up to 2 years.
  Interventions: Procedure: HAIC (Hepatic arterial infusion chemotherapy); Drug: HLX10 (PD-1 antibody); Drug: HLX04 (VEGF antibody)
- HAIC + Placebo (Placebo Comparator): HAIC: FOLFOX, q3w, up to 8 times; Placebo1: saline, iv, q3w, up to 2 years; Placebo2: saline, iv, q3w, up to 2 years.
  Interventions: Procedure: HAIC (Hepatic arterial infusion chemotherapy); Drug: Placebo

INTERVENTIONS:
Procedure: HAIC (Hepatic arterial infusion chemotherapy) — For the HAIC procedure, a 5F catheter was introduced using the Seldinger technique through the femoral artery or the radial artery. Then, angiographic surveys of the celiac trunk and superior mesenteric artery were performed. According to tumor size, location, and arterial supply, the catheter or a 2.7F microcatheter was advanced into the hepatic artery at the level of selective segmental, lobar, or whole liver. The catheter or microcatheter was connected to an external infusion pump. The following regimen of modified FOLFOX was administered: oxaliplatin, 85mg/m2 for 2 hours; leucovorin, 400mg/m2; and 5-fluorouracil, 2400mg/m2 for 44-46 hours. After HAIC treatment, the catheter or microcatheter, and the sheath were removed.
Drug: HLX10 (PD-1 antibody) — PD-1 antibody with proven efficacy in advanced hepatocellular carcinoma
  Arms: HAIC + HLX10 + HLX04
Drug: HLX04 (VEGF antibody) — Combination of PD-1 antibody and VEGF antibody might promote the efficacy of HAIC in hepatocellular carcinoma with major portal vein thrombosis.
  Arms: HAIC + HLX10 + HLX04
Drug: Placebo — Placebo
  Arms: HAIC + Placebo

SUMMARY:
This is a randomized, double-blinded, controlled, phase II study. The purpose is to evaluate efficacy and safety of the combination therapy of HAIC (Hepatic arterial infusion chemotherapy) with HLX10 (PD-1 antibody) and HLX04 (VEGF antibody) compared with HAIC and placebo in patients with hepatocellular carcinoma with major portal vein tumor thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to attend the study and having given the ICF
2. Age ≥18
3. Have a HCC diagnosis confirmed by radiology, histology, or cytology
4. HCC is diagnosed at Barcelona Clinic Liver Cancer (BCLC) Stage C with major portal vein tumor thrombosis ( VP3～4, or Cheng's II～IV)
5. Have not accepted any of systemic therapy for HCC such as systemic chemotherapy, molecular targeted drugs, immunotherapy.
6. At least 1 measurable intrahepatic lesion suitable for repeat assessments according to RECISTv1.1 criteria and it has not undergone surgery, radiology and/or other regional therapy (including but not limited to radiofrequency ablation, percutaneous ethanol injection, freezing therapy, high intensity focused ultrasound, transcatheter arterial chemoembolization, transcatheter arterial embolization). But if it progressed after the regional therapy, it could be selected as a target lesion. The local regional therapy must be done 4 weeks before randomization and the related AEs must recover to ≤ CTCAE grade 1.
7. Child-Pugh score ≤7
8. Eastern Cooperative Oncology Group (ECOG) 0 or 1
9. Expected life time is over 12 weeks.
10. HBV-DNA < 2000 IU/mL
11. Organs function:

Platelet count ≥75×109/L Absolute neutrophil count (ANC) ≥1.5×109 /L White blood cell count ≥3.0×109 /L Haemoglobin ≥9.0 g/dL Serum total bilirubin ≤1.5×ULN ALT ≤5×ULN, and AST ≤5×ULN（ALT ≤3×ULN, and AST ≤3×ULN, if HCV-RNA is detectable） Albumin ≥28 g/L INR ≤1.5×ULN PT ≤1.5×ULN APTT ≤1.5×ULN Creatinine clearance (CL) >50 mL/min or serum creatinine ≤1.5×ULN Urine protein ≤1+ or ≤1.0g/24h 12. Patient is not fertile or willing and able to obey effective contraception.

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinoma and HCC
2. History of hepatic encephalopathy
3. History of GI bleeding within 6 months, or investigator defined with high risk of haemorrhage for esophageal varices
4. With distant metastasis (hilar lymph nodes metastasis is allowed)
5. Co-infection of HBV and HCV
6. History of other malignancy within 5 years except for healed local tumor.
7. History of or plan to accept allogenic organ transplantation
8. Ascites requiring invasive intervention (e.g. paracentesis) to maintain symptomatic control (every month or more often)
9. History of myocardial infarction or unstable angina or uncontrolled arrythmia or stroke or cerebral hemorrhage within 6 months prior to randomization. QTcF value ≥450ms（male）or ≥470ms（female） detected by 12-lead electrocardiogram.
10. New York Heart Association Grade ≥2 congestive heart failure or LVEF <50%
11. Uncontrolled hypertension
12. History of hypertensive crisis or hypertensive encephalopathy
13. Active infection including but not limited to tuberculosis and HIV
14. With interstitial lung disease, lung fibrosis, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia and serious impairment in lung function
15. Active autoimmune disorders except patients with substitutional treatment with thyroid hormone and type I diabetes under treatment with insulin.
16. Receipt of live attenuated vaccine within 28 days prior to randomization
17. Current or prior use of steroids (>10mg/d prednisone) or immunosuppressive medication within 14 days before randomization
18. Significant traumatic injury or major surgical procedure within 28 days prior to randomization
19. Receipt of checkpoint inhibitors or T cell costimulatory drugs
20. Receipt of bevacizumab or its analogues
21. Involved in another clinical trial less than 14 days before randomization
22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
23. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control
24. Active bleeding, with history of ≥grade 3 bleeding within 6 months, or ≥grade 2 bleeding within 3 months
25. Use of anti-thrombotics within 5 days prior to randomization
26. In need of NSAIDs for long-term treatment.
27. With one of the following diseases within 6 months before randomization:

(1) Digestive fistula, perforation and abscess (2) Gastrointestinal obstruction (3) Abdominal infection or inflammation (4) Major vascular disease 28. With severe and green wound, active ulcer or untreated fracture 29. History of drug abuse 30. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to screen for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | The proportion of patients with complete response or partial response, through study completion, an average of 3 years.
  efficacy

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of the first documented progression or date of death from any cause, whichever comes first, up to 48 months
  efficacy
Duration of response | From date of randomization until the date of first documented progression, up to 48 months
  efficacy
Time to response | From date of randomization until the date of first documented response, up to 48 months
  efficacy
Time to progression | From date of randomization until the date of first documented progression, up to 48 months
  efficacy
Overall survival | From date of randomization until death from any cause, up to 48 months
  efficacy
Progression free survival rate at 12-month time point | From date of randomization until 12-month time point
  efficacy
Overall survival rate at 12-month time point | From date of randomization until 12-month time point
  efficacy

OTHER OUTCOMES:
Objective response rate according to iRECIST criteria | The proportion of patients with complete response or partial response according to iRECIST criteria, through study completion, an average of 3 years.
  efficacy
Progression free survival according to iRECIST criteria | From date of randomization until date of confirmed progression according to iRECIST criteria, up to 48 months
  efficacy
Duration of response according to iRECIST criteria | From date of randomization until date of confirmed progression according to iRECIST criteria, up to 48 months
  efficacy
Time to response according to iRECIST criteria | From date of randomization until date of the first documented response according to iRECIST criteria, up to 48 months
  efficacy
Time to progression according to iRECIST criteria | From date of randomization until date of confirmed progression according to iRECIST criteria, up to 48 months.
  efficacy
Adverse events rate | From date of randomization until 30 days after the last treatment or beginning of new anti-cancer therapy, whichever comes first, up to 48 months
  Safety
Severe adverse events rate | From date of randomization until 90 days after the last treatment, up to 48 months
  Safety
Discontinuation rate due to any adverse events | From date of randomization until the last treatment, up to 48 months
  Safety